CLINICAL TRIAL: NCT00427388
Title: Phase IV Study of Perioperative Steroid's Effects on Death or MI in High-Risk Patients Undergoing Cardiac Surgery Requiring Cardiopulmonary Bypass
Brief Title: Steroids In caRdiac Surgery Trial (SIRS Trial)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Richard Whitlock, Assistant Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIRS 2007
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Cardiac Surgical Procedures; Cardiopulmonary Bypass; Systemic Inflammatory Response Syndrome
Keywords: Cardiac Surgical Procedures; Cardiopulmonary Bypass; Systemic inflammatory Response Syndrome; Steroid; Myocardial Infarction; Randomized Clinical Trial
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Myocardial Infarction | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): 500 mg of methylprednisolone divided into two intravenous doses of 250 mg each, one during anesthetic induction and the other on CPB initiation
  Interventions: Drug: Methylprednisolone
- Placebo (Placebo Comparator): 500 mg of matching placebo (normal saline solution) divided into two intravenous doses of 250 mg each, one during anesthetic induction and the other on CPB initiation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — Given by IV in 2 doses (250 mg each dose for a total of 500 mg)
  Arms: Treatment
Other: Placebo — Given in 2 IV doses (approximately 4 ml of 0.9% normal saline solution in each dose)
  Arms: Placebo

SUMMARY:
SIRS trial is a large simple study in which high-risk patients undergoing cardiac surgery requiring the use of cardiopulmonary bypass (CPB) are randomly allocated to receive a pulse dose of Methylprednisolone or a matching placebo. Cardiopulmonary bypass initiates a systemic inflammatory response that facilitates development of post-operative complications. SIRS will confirm or deny the potential clinical benefits of suppressing this response through the use of systemic steroids. Specifically, does 250 mg of intravenous Methylprednisolone given twice, once on anesthetic induction and again on CPB initiation, result in improved early survival and less myocardial infarction in high-risk cardiac surgery patients requiring CPB?

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) is a commonly performed surgical procedure with over 500,000 per year in North America. CPB initiates a systemic inflammatory response characterized by both cell and protein activation. Platelets, neutrophils, monocytes, macrophages, coagulation, fibrinolytic, and kallikrein cascades all take part in what results in increased endothelial permeability, vascular, and parenchymal damage. These inflammatory pathways facilitate development of post-operative complications including thrombosis, myocardial injury and infarction, respiratory failure, renal and neurological dysfunction, bleeding disorders, altered liver function and ultimately, multiple organ failure.

In an attempt to minimize the deleterious effects of CPB, investigators have tested a variety of strategies in cardiac surgery ranging from the complete avoidance of CPB, to the use of biocompatible circuits and pharmacologic agents to abrogate the systemic response. Investigators have consistently demonstrated the efficacy of steroids as the most potent anti-inflammatory agent for use during CPB. In fact, from the available evidence, the 2004 AHA guidelines for coronary artery bypass grafting (CABG) "support liberal prophylactic use in patients undergoing extracorporeal circulation". However, the trials that do exist within this literature are focused on biochemical endpoints and are insufficiently powered to make conclusions on hard clinical endpoints. Our pilot RCT, SIRS I, demonstrated the efficacy of a low dose steroid protocol in the suppression of this inflammatory cascade. We hypothesize that this low dose protocol will yield clinical benefit while avoiding the potential adverse effects of steroids which are known to be dose dependent.

The primary aim of the SIRS trial is to determine if perioperative pulse dose Methylprednisolone results in improved early survival and less myocardial infarction in cardiac surgery requiring CPB. Additional secondary aims of the SIRS trial are to determine the effect of steroids on other clinical outcomes including length of stay, new onset atrial fibrillation, transfusion requirements, infectious, wound, and gastrointestinal complications.

The design of the SIRS trial is a prospective multicentre international double-blind placebo controlled randomized clinical trial. The sample size of 7500 patients will have 80% to 90% power to detect a 20-30% RRR for the primary outcome with an α=0.05 (two-sided), anticipating a 6% rate of death in the control arm. Our aim is to have 85 international centers participate which, recruiting at 5 patients per month, would complete recruitment in 36 months. This will be a large trial with a simple design and objective outcomes.

A sub-group of patients will be enrolled in a renal sub-study. This sub-study will determine if the risk of acute kidney injury is lower in patients treated with intravenous steroid versus placebo, if steroids lead to better preservation of kidney function six months after cardiac surgery, and whether the impact of steroid exposure differs in patients with and without pre-operative chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Require CPB for any cardiac surgical procedure (such as CABG, Valve, Aorta, or combined procedures)
3. Must have a EuroSCORE ≥ 6
4. Provide written informed consent

NOTE: For participating sites in India, China and Hong Kong, the following eligibility criteria will be applied:

1. Age greater than 18 years
2. Require CPB for any cardiac surgical procedure (such as CABG, Valve, Aorta, or combined procedures)
3. Must have at least one of the following:

   1. EuroSCORE greater than or equal to 4 and undergoing valvular surgery
   2. EuroSCORE greater than or equal to 6 and undergoing any other cardiac surgery procedure (i.e. CABG, Aorta)
4. Provide written informed consent

Exclusion Criteria:

1. Use of systemic corticosteroids
2. History of bacterial or fungal infection in last 30 days
3. Allergy/intolerance to corticosteroids
4. Will receive Aprotinin
5. Previous participation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7507 (Actual)
Dates: Start 2007-06; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Mortality at 30 days | 30 days post-randomization
Composite | 30 days post-randomization
  Incidence of the composite outcome of death, myocardial infarction, stroke, renal failure (KDIGO Stage III acute kidney injury, 2012 Kidney Disease Improving Global Outcomes (KDIGO) guidelines), or respiratory failure within 30 days

SECONDARY OUTCOMES:
MI or Mortality at 30 days | 30 days post-randomization
  Composite of death or significant myocardial infarction within 30 days post-randomization
Mortality at 6 months | 6 months post-randomization
  All-cause mortality at 6 months post-randomization
Atrial Fibrillation | 30 days post-randomization
  New onset atrial fibrillation within 30 days post-randomization
Transfusion Requirements | 24 hours post-surgery
  Transfusion requirements within first 24 hours post-operative
Chest Tube Output | 24 hours post-surgery
  Chest tube output within first 24 hours post-operative
ICU and Hospital Length of Stay | Hospital Discharge
  Length of ICU stay and hospital stay
Infection | 30 days post-randomization
  Infection within 30 days post-randomization
Delirium | 3 days post-surgery
  Delirium at day 3 post-operative
Wound Complication | 30 days post-randomization
  Wound complication within 30 days post-randomization
GI Hemorrhage | 30 days post-randomization
  GI hemorrhage or GI perforation within 30 days post-randomization
Insulin Use | 24 hours post-surgery
  Post-operative insulin use within the first 24 hours after surgery
Peak Blood Glucose | 24 hours post-surgery
  Peak blood glucose within the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Salim Yusuf, MD, DPhil, Principal Investigator — Pranic Healing Research Institute; Kevin Teoh, MD, MSc, Principal Investigator — McMaster University; Richard P Whitlock, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Whitlock RP, Young E, Noora J, Farrokhyar F, Blackall M, Teoh KH. Pulse low dose steroids attenuate post-cardiopulmonary bypass SIRS; SIRS I. J Surg Res. 2006 May 15;132(2):188-94. doi: 10.1016/j.jss.2006.02.013. Epub 2006 Mar 29. PMID 16566943
- [Background] Whitlock RP, Rubens FD, Young E, Teoh KH. Pro: Steroids should be used for cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 2005 Apr;19(2):250-4. doi: 10.1053/j.jvca.2005.02.010. No abstract available. PMID 15868539
- [Background] Whitlock R, Teoh K, Vincent J, Devereaux PJ, Lamy A, Paparella D, Zuo Y, Sessler DI, Shah P, Villar JC, Karthikeyan G, Urrutia G, Alvezum A, Zhang X, Abbasi SH, Zheng H, Quantz M, Yared JP, Yu H, Noiseux N, Yusuf S. Rationale and design of the steroids in cardiac surgery trial. Am Heart J. 2014 May;167(5):660-5. doi: 10.1016/j.ahj.2014.01.018. Epub 2014 Mar 1. PMID 24766975
- [Background] Garg AX, Vincent J, Cuerden M, Parikh C, Devereaux PJ, Teoh K, Yusuf S, Hildebrand A, Lamy A, Zuo Y, Sessler DI, Shah P, Abbasi SH, Quantz M, Yared JP, Noiseux N, Tagarakis G, Rochon A, Pogue J, Walsh M, Chan MT, Lamontagne F, Salehiomran A, Whitlock R; SIRS Investigators. Steroids In caRdiac Surgery (SIRS) trial: acute kidney injury substudy protocol of an international randomised controlled trial. BMJ Open. 2014 Mar 5;4(3):e004842. doi: 10.1136/bmjopen-2014-004842. PMID 24598306
- [Derived] Garg AX, Chan MTV, Cuerden MS, Devereaux PJ, Abbasi SH, Hildebrand A, Lamontagne F, Lamy A, Noiseux N, Parikh CR, Perkovic V, Quantz M, Rochon A, Royse A, Sessler DI, Shah PJ, Sontrop JM, Tagarakis GI, Teoh KH, Vincent J, Walsh M, Yared JP, Yusuf S, Whitlock RP; SIRS Investigators. Effect of methylprednisolone on acute kidney injury in patients undergoing cardiac surgery with a cardiopulmonary bypass pump: a randomized controlled trial. CMAJ. 2019 Mar 4;191(9):E247-E256. doi: 10.1503/cmaj.181644. PMID 30833491
- [Derived] Theriault S, Whitlock R, Raman K, Vincent J, Yusuf S, Pare G. Gene Expression Profiles for the Identification of Prevalent Atrial Fibrillation. J Am Heart Assoc. 2017 Jun 30;6(7):e006057. doi: 10.1161/JAHA.117.006057. PMID 28666990
- [Derived] Whitlock RP, Devereaux PJ, Teoh KH, Lamy A, Vincent J, Pogue J, Paparella D, Sessler DI, Karthikeyan G, Villar JC, Zuo Y, Avezum A, Quantz M, Tagarakis GI, Shah PJ, Abbasi SH, Zheng H, Pettit S, Chrolavicius S, Yusuf S; SIRS Investigators. Methylprednisolone in patients undergoing cardiopulmonary bypass (SIRS): a randomised, double-blind, placebo-controlled trial. Lancet. 2015 Sep 26;386(10000):1243-1253. doi: 10.1016/S0140-6736(15)00273-1. PMID 26460660